CLINICAL TRIAL: NCT05468580
Title: Coeliac Artery Release or Sham Operation in Patients Suspected of the Median Arcuate Ligament Syndrome
Brief Title: Coeliac Artery Release or Sham Operation
Acronym: CARoSO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medisch Spectrum Twente (Other)
Collaborators: Medical School Medisch Spectrum Twente (Unknown); Techmed University of Twente (Unknown); Erasmus Medical Centre (Unknown)
Responsible Party: Principal Investigator, R. H. Geelkerken, Principal Investigator, Medisch Spectrum Twente
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: X
Record Dates: First submitted 2022-07-14; First posted 2022-07-21 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Mesenteric Ischemia; Median Arcuate Ligament Syndrome; Dunbar Syndrome; Coeliac Artery Compression; Celiac Artery Compression Syndrome
Keywords: MALS; Mesenteric ischaemia; Quality of Life; Coeliac Artery Release; Sham Operation; Healthcare Costs
MeSH Terms: conditions — Mesenteric Ischemia; Median Arcuate Ligament Syndrome

STUDY DESIGN:
Intervention Model Description: A nationwide randomized placebo-controlled patient and observer blinded clinical superiority trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients are randomized in a 1:1 fashion (stratified on preoperative abdominal pain VAS, psychiatric comorbidities and gender) for either endoscopic Coeliac Artery Release (eCAR) or a sham operation.The randomization takes place in the operating room by a randomization program. Except for the surgical team, all care providers are blinded. To maintain the blinding, there will be no (substantive) contact between the members of the operating team and the patient postoperatively (or in follow up).
  In the event of an emergency in a patient included in the CARoSO study envelopes will be 24/7 available to break the blind. Furthermore the study will be unblinded when the difference in effectiveness as described in the hypothesis is achieved for the primary outcome after the analyses on the 6 months outcomes (both primary and secondary) have been completed for all included subjects. This decision will be made by the Data Safety and Monotoring Board.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endoscopic Coeliac Artery Release (eCAR) (Active Comparator): Patients randomized in the Intervention Group.
  Interventions: Procedure: Endoscopic Coeliac Artery Release (eCAR)
- Sham Operation (Sham Comparator): Patients randomized in the Sham group.
  Interventions: Procedure: Sham Operation

INTERVENTIONS:
Procedure: Endoscopic Coeliac Artery Release (eCAR) — Endoscopic Coeliac Artery Release (eCAR); The Median Arcuate Ligament will be cleaved via an endoscopic retroperitoneal approach using a 4 trocar technique described in detail by van Petersen (12). To rule out learning curves and procedural variation all the procedures will be performed by two experienced eCAR surgeons in the MST-Dutch Expert Centre of Gastrointestinal Ischemia. All procedures will be videotaped. Both eCAR surgeons will not be involved in the follow up procedures.
  Arms: endoscopic Coeliac Artery Release (eCAR)
Procedure: Sham Operation — The sham operation consists of making 4 incisions up to the fascia similar to endoscopic AC release (eCAR). After 60 to 75 minutes of general anesthesia, in accordance with the average operating time of eCAR, the sham operation is ended. This study design allows for patient and observer blinding and for the sham group the eCAR approach is still feasible if the CARoSO outcome support this without applying additional scar tissue.
  Arms: Sham Operation

SUMMARY:
In patients with Median Arcuate Ligament Syndrome (MALS), significant external compression of the coeliac artery (CA) by the median arcuate ligament (MAL) increasing mucosal ischemia (1,2) is assumed to cause chronic disabling postprandial abdominal pain, weight loss, and consequently lethargy and social deprivation (3,8). The majority of these patients have had a long medical journey before the diagnosis MALS is considered resulting in a substantial burden of disease and high healthcare and societal costs.

Although a Systematic Review have shown a sustainable symptom relief of 68% and a significant and durable improvement of quality of life after surgical treatment for MALS (4), there is still no (inter)national consensus on the existence and treatment of MALS (1, 5, 6, 7).

Two recent guidelines (3, 8) concluded that patients with MALS might be considered for surgical CA release (Recommendation 25 GRADE 2D; expert agreement 96%, Terlouw 2020). To end the ongoing debate and to enable the development of evidence-based guidelines for the management of MALS, both guideline committees recommend to perform a blinded, randomised controlled trial comparing a CA release with a sham operation. The proposed Coeliac Artery Release or Sham Operation study will either underline the usefulness of eCAR as a minimal invasive (cost)effective treatment for MALS or it will prohibit a meaningless intervention in patients with disabling abdominal symptoms.

If the CARoSO study proves that the treatment of MALS by eCAR is effective, to 490 patients with chronic disabling abdominal symptoms per year can be treated in the Netherlands. Effective treatment of MALS is expected to result in mean health gain of 6.05 Quality Adjusted Life Years (QALYs)/patient and has the potency to reduce the substantial productivity loss and healthcare consumption caused by MALS, resulting in a saving up to M€4.3/year. The outcome of the CARoSO study will be translated into strong recommendations in the coming updates of the relevant (inter)national multidisciplinary guidelines and will be adapted in daily practice.

DETAILED DESCRIPTION:
The involved professions and the patient representatives unanimously recommend as primary endpoint for this study the proposed disease specific outcome measure: symptom relief measured on a VAS and PGI-I scale. This clinical outcome parameter can be reliable assessed within 6 months after the CA release (1, 9, 10). A two years follow up is suggested to extinguish the positive effect of attention in the diagnostic phase (11).

This study design allows for patient and observer blinding and for the sham group the eCAR approach is still feasible if the CARoSO outcome support this without applying additional scar tissue. A sham operation without skin incisions results in unblinding for the patient and the observer and thus undermines the basis of the evidential value of this study. There are no known cases where irreversible damage such as the intestinal infarction has occurred due to not treating this condition. Possible risks of not treating are continuous (pain) complaints and weight loss. The patients who undergo the sham operation and who still have complaints after unblinding of the study and proven effectivity of eCAR can still undergo the endoscopic AC release.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a consensus diagnosis of MALS based on a multidisciplinary discussion in the two Dutch expert centers for Mesenteric Ischemia (Medisch Spectrum Twente and Erasmus Medical Centre). The multidisciplinary team contains of a vascular surgeon, gastroenterologist, radiologist as recommended in the guidelines.
* Typical complaints: post-prandial pain and at least two of the following: dietary modification, unexplained weight loss, unexplained diarrhea.
* Eccentric stenosis of ≥70% of the AC at the medial arcuatum ligament, demonstrated by two imaging techniques (duplex, MRA, CTA or DSA), including at least an inspiration and expiration CTA with 1mm sections. (Definition percent stenosis according to ECST 1998 formula: % stenosis = (1 - [diameter at the site of stenosis/estimated original diameter at the site of the stenosis]) x 100).
* Ultrasound Abdomen without other more common abnormalities.
* Gastroscopy-duodenoscopy without abnormalities, unless appropriate for mucosal ischemia.

Exclusion Criteria:

* Patient not suitable for endoscopic AC release (e.g. previous surgery in the operating area).
* Pregnancy.
* Previous (endovascular) intervention of the visceral arteries.
* A significant stenosis in the superior or in the inferior mesenteric artery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
The number of patients with significant reduction in abdominal symptoms on a VAS scale | 6 months after randomization
  The change in abdominal symptoms is measured with a composite primary end point (CPE) at 6 months after randomization existing of o the daily visual analogue scale (VAS) for abdominal pain
  * every day for seven days, the patients is asked to indicate the average abdominal pain of the past 24 hours on a VAS, this calculates the average VAS for that week.
  * The PGI-I consists of one question about the change in symptoms compared to before surgery indicated on a 7-point Likert scale with the possible answers: "very much improved", "greatly improved", "somewhat improved", " no change", "slightly deteriorated", "greatly deteriorated" and "very much worse". - A significant reduction in abdominal symptoms at 6 months after randomization is defined as an o a reduction in mean abdominal pain VAS (0-100) of ≥50% compared to baseline
The number of patients with significant reduction in abdominal symptoms. | 6 months after randomization
  The change in abdominal symptoms is measured with a composite primary end point (CPE) at 6 months after randomization o "much improved" or "very much improved" symptoms on the PGI-I (12) (7-point Likert Scale). The PGI-I consists of one question about the change in symptoms compared to before surgery.

SECONDARY OUTCOMES:
Abdominal pain measured with mean abdominal pain VAS endpoint) | Preoperative and 3, 6, 12 and 18 months after operation
  Visual Analogue Scale from 0-100
Change in complaints measured with the PGI-I | 3, 6, 12 and 18 months after operation
  PGI-I on a 7-point Likert Scale
Abdominal pain measured with worst abdominal pain VAS | Preoperative and 3, 6, 12, 18 and 24 months after operation
HR-QoL measured with the EQ-5D-5L | Preoperative and 3, 6, 12, 18 and 24 months after operation
  Visual Analogue Scale from 0-100
HR-QoL measured with the SF-12 | Preoperative and 3, 6, 12, 18 and 24 months after operation
  SF-12 from 0-100
Productivity loss measured with the iPCQ (Productivity Costs Questionnaire) | 3, 6 and 24 months after randomization
  Measured in euro per patient
Healthcare consumption measured with the iMCQ | 3, 6 and 24 months after operation
  Measured in euro per patient
Cost-utility ratio (ICUR) of AC release compared to a sham operation | 3, 6 and 24 months after operation
  Cost per additional QALY in 6 months
The number of anatomically successful procedures, defined as ≤30% stenosis (diameter permeated lumen/diameter artery*100) measured with a CTa/MRa | 6 months after operation
  Amount of anatomically succesful procedures
The number of days until return to a normal diet | 24 months after operation
Weight | Preoperative and 3, 6, 12 and 18 months after operation
  Kilograms
Success of blinding | 3, 6, 12, 18 and 24months after operation
  By asking the patient in which treatment group they were randomzied
Complications classified in the Clavien-Dindo classification | 30 days after operation
  Questionnaire
Percentage of patients undergoing additional PTA or other surgical treatment | 24 months after operation
  Percentage of patients
QoL measured by WHO-QoL Bref | Preoperative and 3, 6, 12, 18 and 24 months after operation
  Scale 0-100

CONTACTS AND LOCATIONS:
Overall Officials: RH Geelkerken, MD PHD, Principal Investigator — Medisch Spectrum Twente
Locations (1):
- Medisch Spectrum Twente, Enschede, Overijssel, Netherlands

REFERENCES:
- [Background] Mensink PB, van Petersen AS, Kolkman JJ, Otte JA, Huisman AB, Geelkerken RH. Gastric exercise tonometry: the key investigation in patients with suspected celiac artery compression syndrome. J Vasc Surg. 2006 Aug;44(2):277-81. doi: 10.1016/j.jvs.2006.03.038. PMID 16890853
- [Background] Berge ST, Safi N, Medhus AW, Sundhagen JO, Hisdal J, Kazmi SSH. Perioperative Microcirculatory Changes Detected with Gastroscopy Assisted Laser Doppler Flowmetry and Visible Light Spectroscopy in Patients with Median Arcuate Ligament Syndrome. Vasc Health Risk Manag. 2020 Aug 10;16:331-341. doi: 10.2147/VHRM.S252192. eCollection 2020. PMID 32982262
- [Background] Bjorck M, Koelemay M, Acosta S, Bastos Goncalves F, Kolbel T, Kolkman JJ, Lees T, Lefevre JH, Menyhei G, Oderich G, Esvs Guidelines Committee, Kolh P, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Kakkos S, Koncar I, Sanddal Lindholt J, Vega de Ceniga M, Vermassen F, Verzini F, Document Reviewers, Geelkerken B, Gloviczki P, Huber T, Naylor R. Editor's Choice - Management of the Diseases of Mesenteric Arteries and Veins: Clinical Practice Guidelines of the European Society of Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2017 Apr;53(4):460-510. doi: 10.1016/j.ejvs.2017.01.010. No abstract available. PMID 28359440
- [Background] Metz FM, Blauw JTM, Brusse-Keizer M, Kolkman JJ, Bruno MJ, Geelkerken RH; Dutch Mesenteric Ischaemia Study Group. Systematic Review of the Efficacy of Treatment for Median Arcuate Ligament Syndrome. Eur J Vasc Endovasc Surg. 2022 Dec;64(6):720-732. doi: 10.1016/j.ejvs.2022.08.033. Epub 2022 Sep 6. PMID 36075541
- [Background] Szilagyi DE, Rian RL, Elliott JP, Smith RF. The celiac artery compression syndrome: does it exist? Surgery. 1972 Dec;72(6):849-63. No abstract available. PMID 5087274
- [Background] Geelkerken RH, van Bockel JH, de Roos WK, Hermans J. Coeliac artery compression syndrome: the effect of decompression. Br J Surg. 1990 Jul;77(7):807-9. doi: 10.1002/bjs.1800770728. PMID 2383757
- [Background] van Dijk LJD, Moons LMG, van Noord D, Moelker A, Verhagen HJM, Bruno MJ, Rouwet EV. Persistent symptom relief after revascularization in patients with single-artery chronic mesenteric ischemia. J Vasc Surg. 2018 Sep;68(3):779-785. doi: 10.1016/j.jvs.2017.12.038. Epub 2018 Mar 6. PMID 29523436
- [Background] Terlouw LG, Moelker A, Abrahamsen J, Acosta S, Bakker OJ, Baumgartner I, Boyer L, Corcos O, van Dijk LJ, Duran M, Geelkerken RH, Illuminati G, Jackson RW, Karkkainen JM, Kolkman JJ, Lonn L, Mazzei MA, Nuzzo A, Pecoraro F, Raupach J, Verhagen HJ, Zech CJ, van Noord D, Bruno MJ. European guidelines on chronic mesenteric ischaemia - joint United European Gastroenterology, European Association for Gastroenterology, Endoscopy and Nutrition, European Society of Gastrointestinal and Abdominal Radiology, Netherlands Association of Hepatogastroenterologists, Hellenic Society of Gastroenterology, Cardiovascular and Interventional Radiological Society of Europe, and Dutch Mesenteric Ischemia Study group clinical guidelines on the diagnosis and treatment of patients with chronic mesenteric ischaemia. United European Gastroenterol J. 2020 May;8(4):371-395. doi: 10.1177/2050640620916681. Epub 2020 Apr 16. PMID 32297566
- [Background] Blauw JTM, Pastoors HAM, Brusse-Keizer M, Beuk RJ, Kolkman JJ, Geelkerken RH, For The Dutch Mesenteric Ischemia Study Group. The Impact of Revascularisation on Quality of Life in Chronic Mesenteric Ischemia. Can J Gastroenterol Hepatol. 2019 Nov 12;2019:7346013. doi: 10.1155/2019/7346013. eCollection 2019. PMID 31781520
- [Background] Metz F, Blauw J, Brusse-Keizer M, Kolkman J, Geelkerken R. Quality of life temporarily improved in patients in whom the diagnosis chronic mesenteric ischemia wasn't confirmed after multidisciplinary evaluation in a tertiary referral centre. Japanese J Gastroenterol Res. 2022;2:1-6.
- [Background] van Petersen AS, Vriens BH, Huisman AB, Kolkman JJ, Geelkerken RH. Retroperitoneal endoscopic release in the management of celiac artery compression syndrome. J Vasc Surg. 2009 Jul;50(1):140-7. doi: 10.1016/j.jvs.2008.12.077. PMID 19563962
- [Background] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145